CLINICAL TRIAL: NCT02500823
Title: Association Between Mitochondrial DNA Copy Number in Peripheral Blood Cells and Risk of Developing Coronary Heart Disease
Brief Title: Association Between Mitochondrial DNA Content and Risk of Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Wenyi Guo, Deputy Director of Department of Cardiovascular Medicine, Air Force Military Medical University, China
Other Study IDs: KY20140813-2
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Heart Disease
Keywords: Mitochondrial DNA copy number; Peripheral blood cells
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Mitochondria are responsible for multiple cellular functions including regulation of energy production, modulation of oxidation-reduction status, generation of reactive oxygen species and apoptosis. Each mitochondrion possesses multiple copies of a mitochondrial genome comprised of independently replicating double stranded DNA (mtDNA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CHD group: 200 consecutive patients were recruited, who have diagnosed with coronary heart disease(CHD) by coronary angiography.
- Control group: The 200 healthy controls without previous CHD history were recruited from individuals who visited investigator's hospital for physical examination during the same time period as the case enrollment.

SUMMARY:
Compelling epidemiological evidence indicates that alterations of mitochondrial DNA, including mutations and abnormal content of mitochondrial DNA (mtDNA), are associated with the initiation and development of cardiovascular disease. This study was undertaken to investigate whether mtDNA copy number in peripheral blood cells could be used as a risk predictor for coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. History of documented myocardial infarction;
2. Prior coronary revascularization intervention (coronary artery bypass graft surgery or percutaneous coronary intervention);
3. The presence of ≥ 50% stenosis in one or more coronary arteries identified during cardiac catheterization;

Exclusion Criteria:

1. History of malignancy or end-stage renal disease;
2. Blood transfusion within one month or prior bone marrow transplantation
3. Patients who reluctant to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 eligible CHD patients were anticipated to include in this study.Moreover, The 200 healthy controls without previous CHD history were also recruited from individuals who visited investigator's hospital for physical examination during the same time period.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Relative copy number of mitochondrial DNA | From date of percutaneous coronary intervention until the date of discharging from hospital, assessed up to 5 days
  The ratio of mitochondrial DNA copy number to hemoglobin copy number was calculated for each sample from standard curves. After that, the ratio for each sample was normalized to a calibrator DNA in order to standardize between different runs, and then defined as the measurement of relative mtDNA copy number.Relative copy number of Mitochondrial DNA were measured in CHD patients in comparison to control group.

CONTACTS AND LOCATIONS:
Overall Officials: WenYi Guo, Professor, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu LP, Cheng K, Ning MA, Li HH, Wang HC, Li F, Chen SY, Qu FL, Guo WY. Association between peripheral blood cells mitochondrial DNA content and severity of coronary heart disease. Atherosclerosis. 2017 Jun;261:105-110. doi: 10.1016/j.atherosclerosis.2017.02.013. Epub 2017 Feb 20. PMID 28242046